CLINICAL TRIAL: NCT03254368
Title: Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging Study of ZGN-1061 in Overweight and Obese Subjects With Type 2 Diabetes Mellitus to Evaluate Glycemic Control, Safety, and Tolerability Over 12 Weeks
Brief Title: Study to Assess the Effects and Safety of ZGN-1061 in Overweight and Obese Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zafgen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZAF-1061-201; U1111-1196-7527 (Registry Identifier: International Clinical Trials Registry Platform)
Record Dates: First submitted 2017-08-07; First posted 2017-08-18 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Type 2 Diabetes Mellitus; Overweight and Obesity
Keywords: Methionine Aminopeptidase 2 Inhibitor; Diabetes Mellitus, Type 2; Blood Glucose; Overweight; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity | interventions — ZGN-1061

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 0.05 mg ZGN-1061 (A) (Experimental): 0.05 mg ZGN-1061 subcutaneous injection once every 3 days
  Interventions: Drug: ZGN-1061
- 0.3 mg ZGN-1061 (B) (Experimental): 0.3 mg ZGN-1061 subcutaneous injection once every 3 days
  Interventions: Drug: ZGN-1061
- 0.9 mg ZGN-1061 (C) (Experimental): 0.9 mg ZGN-1061 subcutaneous injection once every 3 days
  Interventions: Drug: ZGN-1061
- 1.8 mg ZGN-1061 (CC) (Experimental): 1.8 mg ZGN-1061 subcutaneous injection once every 3 days
  Interventions: Drug: ZGN-1061
- Placebo (D) (Placebo Comparator): Placebo subcutaneous injection once every 3 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZGN-1061 — ZGN-1061 is a methionine aminopeptidase 2 inhibitor
  Arms: 0.05 mg ZGN-1061 (A); 0.3 mg ZGN-1061 (B); 0.9 mg ZGN-1061 (C); 1.8 mg ZGN-1061 (CC)
Drug: Placebo — Placebo has the same excipients and appearance as ZGN-1061
  Arms: Placebo (D)

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the study drug ZGN-1061 in participants with type 2 diabetes.

DETAILED DESCRIPTION:
Participants will be enrolled in 1 of 2 groups. Approximately 120 participants will receive 0.05, 0.3, or 0.9 mg of ZGN-1061 or placebo (Group 1). An additional 40 participants will receive 0.9 or 1.8 mg of ZGN-1061 or placebo (Group 2).

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following criteria to participate in this study:

* Be between the ages of 18 and 70 years, inclusive.
* Overweight or obese with a body mass index of at least 27 kg/m².
* Have type 2 diabetes with HbA1c between 7% and 11%.
* For subjects taking approved antidiabetes medications, the doses must be stable as determined by the study doctor.
* For subjects who have had weight-loss surgery (example: gastric banding), the procedure must have occurred at least 1 year ago, and be verified with documentation or by a health professional associated with the surgery.

Exclusion Criteria:

Subjects cannot participate in this research study if they meet any of the following:

* Have taken another study drug or study device within the past 6 months.
* Are taking certain prescribed medications including narcotics or opiates.
* Consistent recent use of insulin.
* Have had recent major surgery or prolonged bed rest, or planning or likely to undergo any surgery during the research study.
* Have a history of bleeding disorders or risk factors for excessive blood clotting.
* Have difficulty giving blood.
* Have a history of drug and/or alcohol abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2018-11-12 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c | 12 weeks
Safety and tolerability as assessed by incidence of adverse events | 12 weeks
Safety and tolerability as assessed by change in medication use, vital signs, physical examination findings, mental well-being questionnaires, laboratory evaluations, and electrocardiogram results | 12 weeks

SECONDARY OUTCOMES:
Change in body weight | 12 weeks
Change in fasting plasma glucose | 12 weeks
Change in insulin | 12 weeks
Change in C-peptide | 12 weeks
Change in proinsulin | 12 weeks
Change in glucagon | 12 weeks
Proportion of subjects achieving HbA1c <7% and ≤6.5% | 12 weeks
Change in beta-cell function | 12 weeks
Change in insulin sensitivity | 12 weeks
Change in preprandial and postprandial glycemic parameters as assessed by a mixed meal tolerance test in a subset of subjects | 12 weeks
Change in waist and hip circumference | 12 weeks
Change in biomarkers relevant to obesity and/or type 2 diabetes | 12 weeks
Change in patient reported outcomes measures | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Kim, MD, Study Chair — Zafgen, Inc.
Locations (23):
- Australia (12):
  - Coffs Harbour GP SuperClinic, Coffs Harbour, New South Wales
  - Northside Health, Coffs Harbour, New South Wales
  - The Aim Centre, Merewether, New South Wales
  - The Boden Institute, Sydney, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Pendlebury Research, Sydney, New South Wales
  - Q-Pharm, Herston, Queensland
  - Griffith University, Gold Coast Campus, Southport, Queensland
  - Southern Adelaide Diabetes & Endocrine Services, Daw Park, South Australia
  - Eastern Clinical Research Unit (ECRU), Box Hill, Victoria
  - Barwon Health, Geelong, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- New Zealand (11):
  - Optimal Clinical Trials, Auckland
  - Middlemore Hospital, Auckland
  - Christchurch Diabetes Centre, Christchurch
  - Southern Clinical Trials, Christchurch
  - Lipid and Diabetes Research Group, Christchurch
  - Clinical Trials New Zealand Ltd, Hamilton
  - P3 Research Hawkes Bay, Hastings
  - P3 Research Wellington, Newtown
  - Lakeland Clinical Trials, Rotorua
  - P3 Research Tauranga, Tauranga
  - Wellington Hospital, Wellington

IPD SHARING:
Plan to Share IPD: No